CLINICAL TRIAL: NCT00033020
Title: Motivational Incentives for Enhanced Drug Abuse Recovery: Methadone Clinics
Brief Title: Motivational Incentives for Enhanced Drug Abuse Recovery: Methadone Clinics. - 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Maxine Stitzer, Ph.D., Johns Hopkins Bayview Medical Center
Organization: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: NIDA-CTN-0007-1; NCT00015418 (obsolete NCT alias)
Record Dates: First submitted 2002-04-05; First posted 2002-04-08 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2010-04

CONDITIONS: Substance-Related Disorders
Keywords: substance use disorders
MeSH Terms: conditions — Substance-Related Disorders | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Behavior Therapy

SUMMARY:
The purpose of this study is to test the utilization of incentive values (considerably lower than those typically used in research clinics) to motivate clients to attend treatment and initiate and sustain abstinence.

DETAILED DESCRIPTION:
The purpose of the proposed research is to implement and systematically evaluate, in community treatment settings, motivational incentive procedures that have been well researched and have proven efficacious in a variety of treatment research clinics. The study will determine if motivational incentives along with standard care therapy is more effective than standard therapy alone for the treatment of patients using cocaine or methamphetamine and entering a substance abuse treatment program.

ELIGIBILITY:
Inclusion Criteria:

1. Recent admission to an opioid substitution (methadone maintenance) CTP. Completed at least 4 weeks of maintenance at time of study entry
2. Evidence of cocaine or methamphetamine use Minimum of one documented positive urine within 2 weeks of study entry. For those exiting a controlled environment, any stimulant use within two weeks of entering the controlled environment

Exclusion Criteria:

1. Unable to give informed consent (fails simple consent quiz)
2. Answers yes to question: Are you in recovery from gambling? That is, have you stopped gambling because of previous gambling problems?

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390
Dates: Start 2001-04; Primary Completion 2003-02 (Actual); Study Completion 2003-02 (Actual)

PRIMARY OUTCOMES:
ASI
Opioid and cocaine use
AIDS risk behavior

CONTACTS AND LOCATIONS:
Overall Officials: Maxine Stitzer, Ph.D., Principal Investigator — Johns Hopkins University
Locations (7):
- United States (7):
  - Aegis Medical Systems, Inc., Bakersfield, California
  - Oasis Clinic, Washington D.C., District of Columbia
  - Glenwood Life Counseling Center, Baltimore, Maryland
  - Lower Eastside Service Center (LESC), New York, New York
  - Greenwich House, Inc., New York, New York
  - ACT, Philadelphia, Pennsylvania
  - Charleston Center, Charleston, South Carolina

REFERENCES:
- See also: Data Elements — http://www.ctndatashare.org/protocol-ctndatashare/new-protocols/nida-ctn-0007